CLINICAL TRIAL: NCT00512798
Title: (Inhibition of NF-kB Signaling in Melanoma Therapy) A Phase I/II Clinical Trial of PS-341, a Proteasome Inhibitor, in Combination With an Extended Continuous Oral Schedule of Temozolomide in Patients With Advanced Refractory Solid Tumors With the Phase II Component Only in Patients With Melanoma
Brief Title: Bortezomib and Temozolomide in Treating Patients With Advanced Refractory Solid Tumors or Melanoma
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: This study was terminated due to lack of efficacy
Sponsor: Vanderbilt-Ingram Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Jeffrey A. Sosman, MD, Professor of Medicine; Director, Melanoma and Tumor Immunotherapy Program; Medical Oncologist, Vanderbilt-Ingram Cancer Center
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VICC PHI 0241; VU-VICC-PHI-0241; VU-VICC-IRB-020510; NCT00209248 (obsolete NCT alias)
Record Dates: First submitted 2007-08-06; First posted 2007-08-08 (Estimated); Results first posted 2012-08-03 (Estimated); Last update posted 2012-10-02 (Estimated); Status verified 2012-09

CONDITIONS: Brain and Central Nervous System Tumors; Melanoma; Solid Tumor
Keywords: stage III melanoma; stage IV melanoma; recurrent melanoma; unspecified adult solid tumor, protocol specific; recurrent adult brain tumor; melanoma (skin)
MeSH Terms: conditions — Central Nervous System Neoplasms; Melanoma; Brain Neoplasms | interventions — Bortezomib; Temozolomide; Immunoenzyme Techniques

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Phase I (Experimental)
  Interventions: Drug: PS-341 (VELCADE); Drug: temozolomide; Other: immunoenzyme technique
- Phase II (Experimental)
  Interventions: Drug: PS-341 (VELCADE); Drug: Temozolomide

INTERVENTIONS:
Drug: PS-341 (VELCADE) — Dose Levels PS-341 (day 1)
  * Level -1 0.7 mg/m2
  * Level 1 1.0 mg/m2
  * Level 2 1.0 mg/m2
  * Level 3 1.3 mg/m2
  * Level 4 1.5 mg/m2
  Other Names: bortezomib
  Arms: Phase I
Drug: temozolomide — Temozolomide (day 8)
  * Level - 1 50 mg/m2
  * Level 1 50 mg/m2
  * Level 2 75/mg/m2
  * Level 3 75 mg/m2
  * Level 4 75 mg/m2
  Other Names: TMZ
  Arms: Phase I
Other: immunoenzyme technique — Not noted
  Other Names: None noted
  Arms: Phase I
Drug: PS-341 (VELCADE) — 1.3 mg/m2 by IV on days 1, 4, 8, and 11 of every 21 days
  Arms: Phase II
Drug: Temozolomide — 75 mg/m2 by mouth, daily, during weeks 2-8 (42 days) of every 9-week course.
  Arms: Phase II

SUMMARY:
RATIONALE: Drugs used in chemotherapy, temozolomide, work in different ways to stop the growth of tumor cells, either by killing the cells or stopping them from dividing. Bortezomib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Giving temozolomide together with bortezomib may kill more tumor cells.

PURPOSE: To determine the best dose of bortezomib and temozolomide and to see how well they work in treating patients with advanced refractory solid tumors or melanoma.

ELIGIBILITY:
Inclusion Criteria - for Phase I

* Histologically proven malignancy (confirmed by Vanderbilt pathologists), advanced non-hematologic malignancy that is not curable by standard surgery, radiation therapy, or chemotherapy. Patients with melanoma, especially those with accessible tumors will be sought for this trial, but this part of the trial will not be limited to only melanoma patients
* No available effective therapy (ie; therapy known to be curative, to prolong survival, to reduce tumor-related symptoms, or to have a tangible, beneficial effect upon the patient)
* Adequate performance status for the study, Eastern Cooperative Oncology Group (ECOG) 0-1
* Adequate baseline organ system function, usually:

  * Absolute neutrophil count > or equal to 1500/uL
  * Hemoglobin > or equal to 9.0g/dL
  * Platelet count > or equal to 100,000/uL
  * Institutional Normalized Ratio (INR) < 1.5 prior to any invasive biopsy of tumor tissue
  * Creatinine < or equal to 1.5x institutional upper limit of normal (IULN) (this may be adjusted for drugs totally dependent upon or independent of renal clearance)
  * Aspartate and alanine aminotransferase < or equal to 2.5x IULN, bilirubin < or equal to 1.5x IULN
* Agreement to use a barrier method of contraception, if potentially fertile
* Ability to understand and willingness to grant informed consent
* Patients with brain metastases are eligible only if the brain lesions are under control for a minimum of 4 weeks, with no progressive symptoms, and off systemic steroids. Patients with primary brain tumors are eligible if their dose of systemic steroids is stable for at least 5 days.
* Completed prior chemotherapy a minimum of 4 weeks previously (6 weeks for BCNU and/or mitomycin C), 4 weeks for prior biologic therapy, and 2 weeks for localized radiation therapy. All treatment related toxicity must have resolved as well. Patients can not receive concomitant radiation therapy
* Patients must be 18 years of age or above and competent to sign an institutionally Institutional Review Board approved informed consent

Exclusion Criteria - for Phase I

* Patients with Grade 2 or greater peripheral neuropathy
* Above a maximum of 320 mg/m2 of CDDP for lifetime previously administered would make patient ineligible. No prior taxanes.
* Uncontrolled or serious infection
* New York Heart Association Class III or IV heart disease or uncontrolled angina
* Myocardial infarction, cerebrovascular accident, or pulmonary embolism within the past 6 months
* Concurrent therapy for cancer
* Inability to comply with protocol-specified procedures (ie, treatment, monitoring, or follow-up)

Inclusion Criteria - for Phase II

* For the phase II trial, all patients must have advanced and incurable melanoma. Disease must be measurable. Histologic proof of disease past the primary site
* No other active malignancy including solid tumors or hematologic cancers within 24 months other than CIS, non-melanoma skin cancer, DCIS of breast, and melanoma in situ
* Melanoma patients can have up to 2 regimens of prior biologic therapies and a single regimen of systemic chemotherapy for disseminated disease.. Chemotherapy is allowed only in the chemotherapy treated patients cohort. Prior TMZ or DTIC is only allowed in those patients enrolled into the prior chemotherapy cohort
* All patients must have ECOG 0-1.
* Adequate baseline organ system function, usually:

  * Absolute neutrophil count > or equal to 1500/uL
  * Hemoglobin > or equal to 9.0g/dL
  * Platelet count > equal to 100,000/uL
  * INR < 1.5 prior to any invasive biopsy of tumor tissue
  * Creatinine < or equal to 1.5x institutional upper limit of normal (IULN) (this may be adjusted for drugs totally dependent upon or independent of renal clearance)
  * Aspartate and alanine aminotransferase < or equal to 2.5x IULN, bilirubin < or equal to 1.5x IULN
* Completed prior chemotherapy a minimum of 4 weeks previously (6 weeks for BCNU and/or mitomycin C), 4 weeks for prior biologic therapy, and 2 weeks for localized radiation therapy. No prior PS-341 is allowed. All treatment related toxicity must have resolved as well. Patients can not receive concomitant radiation therapy. Prior TMZ or DTIC is only allowed in those patients enrolled into the prior chemotherapy cohort
* Patients must be 18 years of age or above and competent to sign an institutionally IRB approved informed consent.

Exclusion criteria - for Phase II

* Patients with Grade 2 or greater peripheral neuropathy.
* Uncontrolled or serious infection requiring parenteral antibiotics
* New York Heart Association Class III or IV heart disease or uncontrolled angina
* Myocardial infarction, cerebrovascular accident, or pulmonary embolism within the past 6 months
* Concurrent therapy for cancer xiii. Inability to comply with protocol-specified procedures (ie, treatment, monitoring, or follow-up)
* Patients with brain metastases are ineligible unless the lesions have been resected or irradiated a minimum of 2 months prior to treatment, be off of steroids, and show no evidence for active disease on MRI,
* Above a maximum of 320 mg/m2 of CDDP for lifetime previously administered would make patient ineligible. No prior taxanes

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2003-06; Primary Completion 2006-07 (Actual); Study Completion 2008-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey A. Sosman, MD, Study Chair — Vanderbilt-Ingram Cancer Center
Locations (1):
- Vanderbilt-Ingram Cancer Center, Nashville, Tennessee, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study remained open to accrual from 6/3/03 to 3/11/08.
Pre-assignment Details: 19 participants were enrolled to the phase I portion of this trial and 28 were enrolled to the phase II portion of this trial. There were also 3 participants that were consented to take part in this trial, but were determined to be ineligible.
Groups:
- Phase I: PS-341 will be administered intravenously at 1.0 mg/m2 of body weight beginning on days 1, 4, 8, and 11 of every 21 days. If toxicity occurs, dose will be lowered to 0.7 mg/m2. Dose can be raised to a maximum of 1.5 mg/m2. Temozolomide will be orally administered daily at 50 mg/m2 of body weight beginning on day 8 for 6 weeks of every 9-week cycle, followed by a 3-week rest. Minimum dose is 50 mg/m2 and maximum dose is 75 mg/m2.
- Phase II: PS-341 and Temozolomide will be administered in the same manner as in Phase I at doses as determined by the Phase I portion of the trial.
Period: Overall Study
Arm/Group | Phase I | Phase II
Started | 19 | 28
Completed | 0 | 1
Not Completed | 19 | 27
Not completed — Death | 0 | 3
Not completed — Adverse Event | 2 | 4
Not completed — Progression of disease | 14 | 20
Not completed — Withdrawal by Subject | 3 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Phase I | Phase II | Total
Number analyzed (Participants) | 19 | 28 | 47
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 15 | 18 | 33
  >=65 years | 4 | 10 | 14
Age Continuous [Median (Full Range); unit: years] | 58 [27 to 74] | 58 [33 to 78] | 58 [27 to 78]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 9 | 13
  Male | 15 | 19 | 34
Region of Enrollment [Number; unit: participants]
  United States | 19 | 28 | 47

OUTCOME MEASURES:

1. Primary Outcome: Optimal Doses of Temozolomide and Bortezomib (Phase I)
Description: The optimal biologic dose (OBD) defined as the dose that achieves the greatest degree of inhibition of NF-κB activation in peripheral blood mononuclear cells when co-administered with Temozolomide
Time Frame: up to 42 days
Population: All Phase I patients who received the study drugs
Measure: Number; unit: mg/m2
Groups:
- Phase I: Patients with advanced, incurable melanoma who are chemotherapy-naive or patients who had undergone prior therapy with Dacarbazine or Temozolomide with treatment failure.
Arm/Group | Phase I
Number analyzed (Participants) | 19
mg/m2
  bortezomib | 1.3
  temozolomide | 75

2. Secondary Outcome: Patients With Inhibition in NF-kB Activation (Phase I)
Description: Patient with a minimum of 50% reduction from baseline on day 8 or day 29 in NF-kB, measured by picograms/milliliter in peripheral mononuclear blood cells
Time Frame: at baseline, on day 8 and on day 29
Population: Phase I patients for whom blood was taken at baseline,on day 8 and on day 29 of each cycle. There was no correlation of change in NF-kB activation with changes in tumor tissue
Measure: Number; unit: participants
Arm/Group | Phase I
Number analyzed (Participants) | 19
participants | 0

3. Secondary Outcome: Patients With Clinical Anti-tumor Activity (Phase I)
Description: Per RECIST criteria v. 1.0: measurable lesions: complete response (CR) disappearance of target lesions, partial response (PR) > 30% decrease in the sum of the longest diameter (LD) of target lesions, progressive disease (PD) > 20% increase in the sum of the LD of target lesions or appearance of new lesions, stable disease (SD) neither sufficient decrease nor increase of the sum of smallest sum of the LD of target lesions
Time Frame: every 9 weeks up to a maximum of 54 weeks
Population: Patients who received treatment and who were available for measurement of lesions.
Measure: Number; unit: participants
Arm/Group | Phase I
Number analyzed (Participants) | 19
participants
  Complete Response | 0
  Partial Response | 4
  Stable Disease | 1
  Progressive Disease | 14

4. Secondary Outcome: Patients With Inhibition of NF-kB (Phase II)
Description: as for outcome 2
Time Frame: at baseline, on day 8 and on day 29
Population: Patients with advanced, incurable melanoma who are chemotherapy-naive and patients who had undergone prior chemotherapy with either Dacarbazine or Temozolomide with treatment failure. No degree of inhibition of NF-kB was observed. Phase II not completed due to lack of efficacy.
Measure: Number; unit: participants
Groups:
- Phase II: Phase II patients who were available for blood draw on the designated days.
Arm/Group | Phase II
Number analyzed (Participants) | 28
participants | 0

5. Primary Outcome: Number of Patients With Clinical Anti-tumor Activity Phase II)
Description: Per RECIST criteria v. 1.0: measurable lesions: complete response (CR) disappearance of target lesions, partial response (PR) > 30% decrease in the sum of the longest diameter (LD) of target lesions, progressive disease (PD) > 20% increase in the sum of the LD of target lesions or appearance of new lesions, stable disease (SD) neither sufficient decrease nor increase of the sum of smallest sum of the LD of target lesions. Patients with CR + PR + SD
Time Frame: every 9 weeks to a maximum of 54 weeks
Population: Patients who were available to measure response to the study drugs.
Measure: Number; unit: participants
Groups:
- Phase II: Patients with advanced, incurable melanoma who are chemotherapy-naive or patients who had undergone prior treatment with Dacarbazine or Temozolomide with treatment failure.
Arm/Group | Phase II
Number analyzed (Participants) | 28
participants
  Complete Response | 0
  Partial Response | 1
  Stable Disease | 5
  Progressive Disease | 22

ADVERSE EVENTS:
Arm/Group | Phase I | Phase II
Serious Adverse Events (participants affected / at risk) | 6/19 | 4/28
Other Adverse Events (participants affected / at risk) | 19/19 | 28/28
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase I (N=19) | Phase II (N=28)
Platelet count decreased (Investigations) | 0 (0) | 1 (1)
Ischemia/infarction (Cardiac disorders) | 0 (0) | 1 (1)
Edema (Cardiac disorders) | 0 (0) | 1 (1)
Thrombosis/embolism (Vascular disorders) | 0 (0) | 1 (1)
Fatigue (General disorders) | 1 (1) | 1 (1)
Wound - infection (Infections and infestations) | 1 (1) | 1 (2)
Nausea (Gastrointestinal disorders) | 1 (1) | 2 (2)
Pancreatitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Muscle weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Death (Gastrointestinal disorders) | 0 (0) | 2 (2)
hemoglobin (Investigations) | 1 (1) | 0 (0)
conduction abnormality/atrioventricular heart block (Cardiac disorders) | 1 (1) | 0 (0)
vomiting (Gastrointestinal disorders) | 1 (1) | 1 (1)
hyperkalemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
depressed level of consciousness (Nervous system disorders) | 1 (1) | 0 (0)
pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
right groin pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
fever (General disorders) | 0 (0) | 1 (1)
creatinine (Investigations) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase I (N=19) | Phase II (N=28)
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 2 (11) | 1 (12)
abdominal pain or cramping (Gastrointestinal disorders) | 8 (57) | 5 (11)
alkaline phosphatase (Investigations) | 3 (22) | 1 (4)
allergic reaction/hypersensivity (Immune system disorders) | 1 (1) | 0 (0)
anorexia (Metabolism and nutrition disorders) | 14 (159) | 12 (83)
apnea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 5 (52) | 5 (33)
arthritis (Musculoskeletal and connective tissue disorders) | 1 (11) | 1 (4)
Ataxia (Nervous system disorders) | 1 (4) | 0 (0)
bone pain (Musculoskeletal and connective tissue disorders) | 3 (10) | 1 (3)
Chest pain (Cardiac disorders) | 2 (12) | 0 (0)
circulatory or cardiac other (Cardiac disorders) | 1 (1) | 0 (0)
conjunctivitis (Eye disorders) | 1 (2) | 0 (0)
constipation (Gastrointestinal disorders) | 13 (103) | 9 (48)
Constitutional symptoms Other (General disorders) | 4 (10) | 1 (7)
Creatinine (Investigations) | 1 (1) | 1 (4)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 2 (4)
Diarrhea patients without colostomy (Gastrointestinal disorders) | 7 (25) | 11 (31)
Dizziness/lightheadedness (Nervous system disorders) | 6 (33) | 3 (15)
Dry skin (Skin and subcutaneous tissue disorders) | 1 (6) | 0 (0)
Dyspepsia/heartburn (Gastrointestinal disorders) | 3 (53) | 8 (38)
Dysphagia, esophagitis, odynophagia (Gastrointestinal disorders) | 2 (3) | 1 (14)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 6 (71) | 9 (27)
Edema (General disorders) | 5 (63) | 8 (124)
Endocrine other (Endocrine disorders) | 0 (0) | 2 (14)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0)
Fatigue (General disorders) | 18 (241) | 24 (234)
Fever (General disorders) | 5 (14) | 5 (30)
GI other (Gastrointestinal disorders) | 6 (66) | 2 (18)
Headache (Nervous system disorders) | 9 (44) | 4 (7)
Hemoglobin (Investigations) | 19 (150) | 22 (199)
Hemorrhage/bleeding with grade 3 or 4 thrombocytopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Hemorrhage/bleeding without grade 3 or 4 thrombocytopenia (Blood and lymphatic system disorders) | 1 (2) | 0 (0)
Hepatic pain (Hepatobiliary disorders) | 1 (1) | 0 (0)
Hypercholesterolemia (Investigations) | 0 (0) | 4 (30)
Hyperglycemia (Metabolism and nutrition disorders) | 2 (5) | 12 (76)
Hyperkalemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypermagnesemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 2 (15) | 9 (76)
Hyperuricemia (Metabolism and nutrition disorders) | 0 (0) | 4 (24)
Hypoglycemia (Metabolism and nutrition disorders) | 0 (0) | 3 (27)
hypocalcemia (Metabolism and nutrition disorders) | 1 (3) | 0 (0)
hypokalemia (Metabolism and nutrition disorders) | 1 (1) | 5 (16)
Hypomagnesemia (Metabolism and nutrition disorders) | 1 (5) | 3 (7)
Hyponatremia (Metabolism and nutrition disorders) | 4 (18) | 7 (37)
Hypotension (Vascular disorders) | 4 (9) | 0 (0)
Infection without neutropenia (Infections and infestations) | 1 (2) | 4 (9)
Insomnia (Psychiatric disorders) | 3 (28) | 7 (34)
Joint, muscle, bone Other (Musculoskeletal and connective tissue disorders) | 3 (34) | 0 (0)
Leukocytes (Blood and lymphatic system disorders) | 4 (15) | 2 (6)
Memory loss (Nervous system disorders) | 0 (0) | 2 (18)
Mood alteration - depression (Psychiatric disorders) | 3 (34) | 7 (45)
Mood alteration - anxiety, agitation (Psychiatric disorders) | 1 (1) | 3 (26)
Mucositis (Gastrointestinal disorders) | 1 (8) | 2 (4)
Muscle weakness (Metabolism and nutrition disorders) | 0 (0) | 3 (28)
Myalgia (Musculoskeletal and connective tissue disorders) | 6 (61) | 3 (25)
Nausea (Gastrointestinal disorders) | 13 (123) | 23 (146)
Neurologic Other (Nervous system disorders) | 2 (18) | 0 (0)
Neuropathy - motor (Nervous system disorders) | 1 (2) | 0 (0)
Neuropathy - sensory (Nervous system disorders) | 5 (107) | 12 (178)
Neutrophils/granulocytes (Investigations) | 2 (7) | 0 (0)
Occular Other (Eye disorders) | 3 (19) | 0 (0)
Pain Other (General disorders) | 11 (150) | 6 (43)
Palpitations (Cardiac disorders) | 2 (4) | 0 (0)
pigmentation changes (Skin and subcutaneous tissue disorders) | 1 (12) | 0 (0)
Platelets (Investigations) | 7 (30) | 9 (79)
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 1 (5) | 0 (0)
Pruritis (Skin and subcutaneous tissue disorders) | 2 (12) | 3 (11)
Pulmonary Other (Respiratory, thoracic and mediastinal disorders) | 2 (24) | 0 (0)
Radiation dermatitis (Injury, poisoning and procedural complications) | 1 (8) | 0 (0)
Rash/desquamation (Skin and subcutaneous tissue disorders) | 7 (45) | 10 (45)
Renal/Genitourinary Other (Renal and urinary disorders) | 2 (3) | 2 (4)
Rigor, chills (General disorders) | 2 (3) | 0 (0)
Sense of smell (General disorders) | 1 (8) | 0 (0)
SGOT (AST) (Investigations) | 3 (18) | 4 (13)
SGPT (ALT) (Investigations) | 3 (16) | 4 (18)
Sinus tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Skin Other (Skin and subcutaneous tissue disorders) | 5 (27) | 2 (12)
Stomatitis/phyaryngitis (Infections and infestations) | 2 (3) | 0 (0)
Supraventricular arrhythmias (Cardiac disorders) | 0 (0) | 2 (14)
Sweating (Skin and subcutaneous tissue disorders) | 6 (48) | 3 (29)
Taste disturbance (General disorders) | 2 (10) | 2 (9)
Tumor Pain (General disorders) | 3 (37) | 11 (80)
Urinary frequency/urgency (Renal and urinary disorders) | 2 (30) | 2 (17)
Vision/blurred vision (Eye disorders) | 1 (3) | 0 (0)
Voice changes/stridor/layrynx (Respiratory, thoracic and mediastinal disorders) | 2 (11) | 0 (0)
Vomiting (Gastrointestinal disorders) | 12 (56) | 14 (54)
Weight gain (Investigations) | 1 (2) | 0 (0)
Weight loss (Investigations) | 0 (0) | 4 (24)
Wound infection (Infections and infestations) | 1 (1) | 4 (12)
Wound non-infectious (Infections and infestations) | 0 (0) | 2 (6)
Cough (Respiratory, thoracic and mediastinal disorders) | 7 (65) | 6 (18)
bruising (Injury, poisoning and procedural complications) | 2 (6) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes